CLINICAL TRIAL: NCT00571103
Title: Open Label, Flexible Dose 12-Week Clinical Trial of the Safety and Efficacy of Acamprosate in the Treatment of Pathological Gambling
Brief Title: Acamprosate in the Treatment of Pathological Gambling
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Iowa (Other)
Collaborators: University of Nebraska (Other); Forest Laboratories (Industry)
Responsible Party: Principal Investigator, Donald Black, Principal Investigator, University of Iowa
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 200608747
Record Dates: First submitted 2007-12-10; First posted 2007-12-11 (Estimated); Results first posted 2017-05-25 (Actual); Last update posted 2017-05-25 (Actual); Status verified 2017-04

CONDITIONS: Pathological Gambling
Keywords: acamprosate, impulse-control disorders
MeSH Terms: conditions — Gambling; Disruptive, Impulse Control, and Conduct Disorders | interventions — Acamprosate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 Open Label (Experimental): Open Label. At visit 2, all participants were started on Acamprosate, 1,998 mg divided into 3 equal doses.
  Interventions: Drug: acamprosate

INTERVENTIONS:
Drug: acamprosate — Two 333mg tablets taken three times daily.
  Other Names: Campral

SUMMARY:
The purpose of this study is to see whether acamprosate (Campral) will curb the desire to gamble in people with pathological gambling disorder.

DETAILED DESCRIPTION:
Because the opiate antagonists appear to be effective in the treatment of pathological gambling (PG), it is reasonable to ask whether acamprosate (calcium acetylhomotaurine; Campral), also FDA approved for the treatment of alcoholism, can be used effectively to treat PG. Acamprosate is not an opioid antagonist; rather, it is assumed that its therapeutic effects are due to actions on GABA receptors. Acamprosate is structurally related to 1-glutamic, which is an excitatory neurotransmitter. It has been proposed that acamprosate decreases the effects of the naturally-occuring excitatory neurotransmitter glutamate in the body. Because chronic alcohol consumption disrupts this system, and the changes last many months after alcohol ingestion is stopped, it is possible that acamprosate restores the glutamate system towards normal. Regardless, acamprosate decreases the pleasant "high" associated with alcohol consumption, and thus decreases the frequency of relapse during abstinence. We hypothesize that acamprosate will have similar actions in persons with PG.

ELIGIBILITY:
Inclusion Criteria:

* Patients will meet DSM-IV (Diagnostic and Statistical Manual 4th Edition) criteria for Pathological Gambling Disorder
* Patients will achieve a SOGS (South Oaks Gambling Screen) score greater than or equal to 5
* Patients will be 18 years old or older
* Patients will speak standard English
* Patients will be able to give written Informed Consent
* Patients will be able to understand and cooperate with study procedures

Exclusion Criteria:

* Patients having a current (past 3 months) substance use disorder (except dependence)
* Patients having a Hamilton Depression Rating score of greater than or equal to 18 or a score on #1 (depressed mood) greater than 1.
* Patients having a clinically significant medical illness
* Patients at risk for aggressive or suicidal behavior
* Patients who have received the following interventions within the proscribed time prior to study entry: 1) a monoamine oxidase inhibitor within the previous 21 days; 2) long-acting phenothiazines within the previous 3 months; 3) other psychotropic drugs within the previous 14 days; 4) flu- oxetine within the previous 4 weeks.
* Patients having severe antisocial or borderline personality disorder
* Patients with a past or current diagnosis of schizophrenia, schizoaffective disorder, psychotic disorder, bipolar disorder, or delirium, dementia, or other clinically significant cognitive disorder.
* Patients initiating individual, group, or couple psychotherapy during the three moths prior to study entry (excluding Gambler's Anonymous)
* Patients having prior exposure to acamprosate

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2007-10; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donald W Black, MD, Principal Investigator — The University of Iowa Carver College of Medicine; Dennis P McNeilly, PsyD, Principal Investigator — University of Nebraska

IPD SHARING:
Plan to Share IPD: No
We do not plan to share individual participant data.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited through newspaper advertising, word of mouth, and lab registries. Subjects were seen in each doctor's clinic respectively.
Pre-assignment Details: Two subjects failed to meet study criteria (their severity of gambling was too low)and 6 subjects were lost to follow-up after the screening visit (Visit One).
Groups:
- Open Label: All subjects received the drug.
Period: Overall Study
Arm/Group | Open Label
Started | 28
Completed | 26 (Of the 28 participants, 1 subject withdrew and 1 was lost to follow-up after their baseline visit.)
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Open Label
Number analyzed (Participants) | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 28
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.0 (16.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 12
Region of Enrollment [Number; unit: participants]
  United States | 28

OUTCOME MEASURES:

1. Secondary Outcome: The Secondary Efficacy Evaluations Will Include the G-SAS (Gambling Symptom Assessment Scale), Clinical Global Impression - Improvement Scale (CGI-I) , and the CGI-S Clinical Global Impression - Severity Scale.
Description: The G-SAS is a 12 item self-report instrument that reflects the subjects urges to gamble and the subjects gambling behavior. Each item is scored on a 5-point scale from 0 (no symptoms) to 4 (extreme symptoms) with a total score range from 0 to 48. The CGI-I is a 7 point scale requiring the clinician to assess how much the patient's illness has improved or worsened relative to a baseline state as: 1, very much improved; 2, much improved; 3, minimally improved; 4, no change; 5, minimally worse; 6, much worse; or 7, very much worse. The CGI-S is a 7-point scale that requires the clinician to rate the severity of the patient's illness at the time of assessment. A patient is assessed on severity of mental illness at the time of rating 1, normal, not at all ill; 2, borderline mentally ill; 3, mildly ill; 4, moderately ill; 5, markedly ill; 6, severely ill; and 7, among the most extremely ill patients.
Time Frame: 8 weeks minus baseline
Population: A total of 39 participants were screened by phone and 5 failed to meet screening criteria and were excluded; 6 did not return for the baseline visit because of follow-up loss or choosing to discontinue participation. of the remaining 28 patients, 1 discontinued and another was lost to follow-up after the baseline visit. That left 26 subjects.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Open Label
Number analyzed (Participants) | 26
units on a scale
  G-SAS | -1.117 (.228)
  CGI-I | -.145 (.031)
  CGI-S | -.199 (.035)

2. Primary Outcome: The Primary Efficacy Measure Was the Yale-Brown Obsessive Compulsive Scale Modified for PG (YBOCS-PG).
Description: The YBOCS-PG (Yale Brown Obsessive Compulsive Scale modified for Pathological Gambling) is used to assess the range and severity of PG symptoms. The scale is a modification of the YBOCS originally developed by Goodman et al. (1989) for use in rating severity and change in subjects with Obsessive Compulsive Disorder. This adaptation is a 10-item clinician-rated questionnaire, which rates (on a 5-point scale from 0 to 4) time spent, distress, interference, resistance, and control in relation to PG urges and behaviors. The scale ranges from 0 to 40 with a higher score representing increased severity in PG.
Time Frame: 8 weeks minus baseline
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Open Label
Number analyzed (Participants) | 26
units on a scale | -.985 (.158)
Statistical Analysis 1: Comparison: Open Label; Test type: Superiority or Other; p = 0.05, Linear mixed effects; Mean Slope = -.985, 95% CI 2-sided [-1 to 1], Standard Error of Mean .158

ADVERSE EVENTS:
Time Frame: Adverse events were collected for eight weeks.
Arm/Group | Open Label
Serious Adverse Events (participants affected / at risk) | 0/28
Other Adverse Events (participants affected / at risk) | 0/28

LIMITATIONS AND CAVEATS:
The sample was relatively small, and there was no comparison group; therefore, our results could have resulted from the placebo effect. Another limitation is the relatively short length of the trial. Furthermore, there were few minority subjects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No